CLINICAL TRIAL: NCT06336265
Title: Clinical Study of Diaphragmatic Ultrasound to Predict the Therapeutic Effect of High Flow Oxygen Therapy in Mild and Moderate Acute Hypoxic Respiratory Failure
Brief Title: Diaphragmatic Ultrasound to Predict the Therapeutic Effect of High-flow Nasal Cannula Oxygen Therapy
Status: Not yet recruiting | Type: Observational
Sponsor: Xingui Dai (Other)
Responsible Party: Sponsor-Investigator, Xingui Dai, Chief Physician, First People's Hospital of Chenzhou
Organization: First People's Hospital of Chenzhou (Other)
Other Study IDs: Diaphragm ultrasound
Record Dates: First submitted 2024-03-13; First posted 2024-03-28 (Actual); Last update posted 2024-03-28 (Actual); Status verified 2024-03

CONDITIONS: Hypoxic Respiratory Failure

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Diaphragm ultrasound — Respiratory parameters, diaphragmatic activity, and variation rate of diaphragmatic thickness were recorded at the beginning of high-flow nasal cannula oxygen therapy, 1 hour after treatment, 3 hours after treatment, 6 hours after treatment, 9 hours after treatment, and 12 hours after treatment.

SUMMARY:
Follow-up was conducted for every patient requiring high-flow nasal cannula oxygen therapy in district 1 of the Intensive Care Department of Chenzhou NO.1 People's Hospital. Patients who met the inclusion criteria but did not meet the exclusion criteria were included for observation. Respiratory parameters, diaphragmatic activity, and variation rate of diaphragmatic thickness were recorded at the beginning of high-flow nasal cannula oxygen therapy, 1 hour after treatment, 3 hours after treatment, 6 hours after treatment, 9 hours after treatment, and 12 hours after treatment. Throughout the procedure, a panel of experts assessed whether the patient needed endotracheal intubation; If yes, the study was terminated; if no, high-flow nasal cannula oxygen therapy was continued, and observation and evaluation were continued until the end point of the study (12 hours after treatment). If patients or their family members do not want to continue to participate in the study during the study, they will be considered as withdrawal. If patients suffer from sudden malignant arrhythmia or cardiac arrest during the study, resulting in death or transfer to other hospitals or other departments during the study, patients will be excluded. Data from dropped and excluded patients were not included in the final statistical analysis. After the data of 269 patients were collected, the study was concluded, and the results and conclusions were derived by statistical analysis.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years old, less than 75 years old,BMI≥18.5kg/m2
2. Mild to moderate type I respiratory failure (100mmHg< PaO2/FiO2≤300mmHg)
3. Mild ventilation dysfunction (pH≥7.3)
4. Mild respiratory distress (respiratory rate > 24 times/min)
5. High-flow nasal cannula oxygen therapy is required
6. The patient and immediate family members agree and sign a written informed consent.

Exclusion Criteria:

1. Patients with severe type II respiratory failure, severe asthma and massive hemoptysis
2. Moderate to severe consciousness disorder, GCS score ≤12 points
3. Cardiogenic pulmonary edema and cardiogenic dyspnea caused by heart failure, heart valvular disease, myocarditis, etc
4. Hemodynamic instability, SBP< 90mmHg, or MAP<65mmHg
5. BMI < 18.5kg/m2
6. Nasal bleeding, nasal space occupying lesions, etc., can not be high-flow nasal cannula oxygen therapy through the nose or nasal obstruction
7. Patients with severe hypoxemia, severe ARDS and other conditions requiring immediate tracheal intubation
8. The patient or family member refuses to participate or does not agree to sign the written informed consent
9. The patient has participated in other research projects with interventions

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with mild to moderate hypoxic respiratory failure who are over 18 years old and less than 75 years old and who do not have serious cardiopulmonary disease, malnutrition, or respiratory obstruction and require high-flow nasal cannula oxygen therapy
Sampling Method: Non-Probability Sample
Enrollment: 269 (Estimated)
Dates: Start 2024-04-01 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Thickness and thickening fraction of Diaphragm | 0-12 hours
  Diaphragm thickness and thickening fraction (TFdi) were measured using a high-frequency linear array probe at the midaxillary line. TFdi = (diaphragm thickness at the end of inspirations - diaphragm thickness at the end of expirations)/diaphragm thickness at the end of expirations × 100%
Diaphragmatic excursion | 0-12 hours
  Diaphragmatic excursion was measured using a low-frequency curved array (" abdomen ") probe located directly below the costal arch on the midline of the clavicle.
Respiratory rate | 0-12 hours
  Respiratory rate of the patient after high-flow nasal oxygen therapy
Incidence of tracheal intubation | 0-12 hours
  After the patient uses high-flow nasal oxygen therapy, the panel determine whether the patient needs to undergo tracheal intubation according to the indicators such as symptoms and signs of the patient.

IPD SHARING:
Plan to Share IPD: No